CLINICAL TRIAL: NCT05618574
Title: Nitrite Supplementation to Mitigate Fatigability and Increase Function in Long COVID Patients
Brief Title: Nitrite Supplementation in Long COVID Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F4409-P; 1I21RX004409 (NIH)
Record Dates: First submitted 2022-11-14; First posted 2022-11-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Long COVID; Cardiorespiratory Fitness
Keywords: Nitrate therapeutics; Long COVID; Skeletal Muscle Mitochondrial Respiration; Fatigability; Cardiorespiratory Fitness
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: In a randomized controlled, blinded design, participants will receive 140 ml per day of Beet-It nitrate beverage (James White Drinks Ltd., Ipswich, UK) for 14 days versus a 210 ml of nitrate-depleted placebo. All participants are encouraged to participate in the standard physical therapy program in the Long COVID clinic 2-3 times per week based on tolerance for activity and recovery needed after each session.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After a participant agrees to consent, their group placement is randomly determined using high quality pseudo-random deviate generator in SAS. Participants in both groups will receive either 140 ml per day of Beet-It nitrate beverage (James White Drinks Ltd., Ipswich, UK) for 14 days versus a 210 ml of nitrate depleted placebo depending on their group placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beet-It nitrate beverage (Active Comparator): Participant will receive 140 ml per day of Beet-It nitrate beverage for for 14 days. All participants will be encouraged to undergo physical therapy 2-3 times per week based on tolerance for activity and recovery needed after each session. Physical therapy will be standardized to include strength, balance, inspiratory muscle training, and aerobic training.
  Participants randomized to this arm will be assessed at baseline and follow-up visits on all outcome measures.
  Interventions: Dietary Supplement: 140 ml per day of Beet-It nitrate beverage (James White Drinks Ltd., Ipswich, UK)
- Nitrate-depleted placebo (Placebo Comparator): Participants will receive 210 ml of nitrate-depleted placebo for 14 days. All participants will be encouraged to undergo physical therapy 2-3 times per week based on tolerance for activity and recovery needed after each session. Physical therapy will be standardized to include strength, balance, inspiratory muscle training, and aerobic training.
  Participants randomized to this arm will be assessed at baseline and follow-up visits on all outcome measures.
  Interventions: Dietary Supplement: 210 ml of nitrate-depleted placebo

INTERVENTIONS:
Dietary Supplement: 140 ml per day of Beet-It nitrate beverage (James White Drinks Ltd., Ipswich, UK) — The investigators propose to study the benefits nitrite therapeutics, using nitrate-rich beetroot juice to increase serum nitrite. The investigators hypothesize that increased nitrite will improve functional metrics and reduce fatigability in Veterans with long COVID as a result of enhanced skeletal muscle mitochondrial respiration. Participant will receive 140 ml per day of Beet-It nitrate beverage for 16 mmol of nitrate/day for 14 days vs the placebo.
  Arms: Beet-It nitrate beverage
Dietary Supplement: 210 ml of nitrate-depleted placebo — Participants randomized to the placebo arm will receive 210 ml of nitrate-depleted beverage (cranberry juice) per day for 14 days.
  Arms: Nitrate-depleted placebo

SUMMARY:
Potential benefits of a nitrate-rich juice supplement to improve skeletal muscle function and associated physical capacity will be studied in patients with Long COVID. Consenting patients with Long-COVID will be randomized to receive Beet-It nitrate beverage group versus a nitrate-depleted placebo beverage. Both groups will receive physical therapy at the long COVID Clinic at VAPHS with therapeutic goals to improve strength, balance, inspiratory, and aerobic capabilities. Physical therapy will last for 2 weeks and include 2 or 3 sessions with a physical therapist a week depending on each individual's exercise tolerance. These sessions can take place on-site or at home (or a hybrid combination) All participants will undergo functional assessments and tissue assessments before and after the 14-day study intervention.

DETAILED DESCRIPTION:
In a proof of concept pilot, the investigators will study 30 Veterans with long COVID, comparing 15 who consume two weeks of daily nitrate-rich beetroot juice versus matched Veterans who consume a nitrate-depleted placebo. Nitrate is metabolized to increase cellular nitric oxide once it is ingested. Nitric oxide (NO) is a signaling molecule that contributes to numerous physiological functions, including enhanced skeletal muscle mitochondrial respiration, which may thereby lead to decreased fatigability and increased physical function. NO is commonly produced from the conversion of the amino acid L-arginine to L-citrulline in the presence of oxygen. However, inorganic nitrate provided as a dietary supplement can serve as an additional substrate for bioactive nitrite and downstream NO, particularly during the ischemic stress of exercise. In this study, consenting patients with Long-COVID will be randomized to receive Beet-It nitrate beverage group as a source of inorganic nitrites and NO, versus a nitrate-depleted placebo beverage. Both groups will undergo simultaneous physical therapy. Primary endpoints center on meaningful clinical changes, including fatigability (i.e., rating of perceived exertion during steady-state walking), cardiorespiratory fitness (i.e., peak oxygen utilization [VO2] as well as submaximal VO2 at anaerobic threshold [VAT]). In addition, serology and skeletal muscle assessments will include nitrate and nitrite levels and mitochondrial respiration to analyze nitrite-mediated mechanisms underlying functional changes.

Principal investigator Daniel Forman, MD has developed expertise in nitrite therapeutics using nitrite capsule supplements for older sedentary adults in relation to sedentariness and heart failure. This SPiRE proposal focuses nitrite therapeutics to both younger and older adults with long COVID.

Aims: We will conduct a pilot randomized controlled trial to study the benefits of nitrate-rich beetroot juice versus placebo in 30 Veterans with a diagnosis of Long COVID. All participants will receive a daily study juice intervention for 2 weeks. All participants will be encouraged to participate in the standard physical therapy program in the Long COVID clinic.

Aim 1: To study the efficacy of nitrate-rich juice supplementation to reduce fatigability as measured by rating of perceived exertion (RPE) during submaximal steady-state 1.5 mile per hour walking after two weeks of treatment in patients with Long Covid. Walking efficiency (VO2 per kg) will also be assessed in association with fatigability.

Aim 2: To study the benefits of nitrate-rich juice supplementation to increase cardiorespiratory fitness (peak oxygen utilization [VO2], VO2 at anaerobic threshold (VAT), 400-meter corridor walk (400MCW), short physical performance battery (SPPB) in patients with Long COVID after two weeks of treatment.

Aim 3: To explore the utility of nitrate-rich juice supplementation to enhance skeletal muscle mitochondrial respiration in patients with Long COVID as measured by ex vivo Oroboros analysis.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with prior COVID-19, with residual symptoms of long COVID including increased fatigability.
* Inclusion limited to age 18 and over

Exclusion Criteria:

* Blood pressure <110/60 mmHg, either systolic or diastolic value which may affect participant safety during assessments will be at the discretion of the study physician
* Unable to hold warfarin, novel oral anticoagulants (NOACs) or aspirin for 3 days prior to muscle biopsy, or to hold thienopyridine medications for 5 days prior to muscle biopsy
* Current use of organic nitrates or phosphodiesterase type 5 (PDE5) inhibitors
* Orthopedic or other chronic condition which limits physical activity or functional testing assessments
* End-stage disease
* Dementia or other reason unable to give informed consent
* Anemia (hemoglobin <11.0 g/dL in men or hemoglobin <10.0 g/dL in women)
* Unstable psychiatric diagnosis
* Clinically significant alcohol intake or substance abuse
* Chronic use of oral corticosteroids or medications that affect muscle function
* Use of anti-bacterial mouthwash or antacids that confound the nitrate/nitrite/NO pathway.
* Suicidal ideations
* Unwilling to hold Viagra-like drugs (i.e. Viagra, Cialis, Levitra, other phosphodiesterase inhibitors)
* Involved in another greater than minimal risk study
* Other clinically unstable medical condition as determined by the study physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Fatigability | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  Rating of Rate of Perceived Exertion (RPE) during the 5th minute of a 5-min of a 1.5 mile per hour steady-state treadmill walking test is used as an assessment of fatigability. RPE scale is from 6 (no physical exertion) - 20 (maximal exertion/very hard).
Walking Efficiency | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  Walking efficiency (VO2/kg) is assessed by incorporating VO2 assessments during the 5-min steady-state walking protocol. This is assessed using cardiopulmonary exercise testing (CPET) equipment. A lower VO2 for the same functional workload indicates improved efficiency.

SECONDARY OUTCOMES:
400m Corridor Walk Test (400MCW) | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  This test measures the amount of time it takes the participant to walk a 400-meter course to assess cardiovascular and pulmonary fitness or to predict adverse outcomes such as mobility disability.
Short Performance Physical Battery (SPPB) | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  The SPPB is a test of balance, gait, strength, and endurance that combines gait speed, chair stand and balance tests. SPPB scaled score ranges from 0 - 12. Scores of 0 indicate that the participant is unable/barely able to perform the tasks, while 12 indicates they completed all tasks optimally.
Mitochondrial Respiration | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  To determine the impact of nitrite-rich juice supplementation on skeletal muscle mitochondrial respiration on patients with Long COVID, muscle biopsy of the vastus lateralis will be completed at baseline and following 2 weeks of supplementation. At each time point muscle respiratory capacity will be measured using the Oroboros-2k system. The main outcome will be state 3 respiration (maxOXPHOS, pmol/mg/min wet.wt.). Data will be reported as Mean +/- standard deviation.
Peak oxygen utilization (VO2) non-normalized | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  Peak VO2 (ml/min) non-normalized to weight will be collected using symptom-limited cardiopulmonary exercise testing (CPET).
VO2 at anaerobic threshold (AT) non-normalized | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  VO2 (ml/min) non-normalized at AT will be assessed using symptom-limited CPET. The VO2 at AT for the general population occurs at approximately 50-60% of the peak VO2.
Veterans RAND-12 (VR-12) | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  The Veterans RAND-12 (VR-12) is a brief, multi-use, self-administered health survey comprised of 12 items. The instrument is primarily used to measure health related quality of life, to estimate disease burden, and to evaluate disease-specific benchmarks. There are two score components: a Physical Component Score a Mental Component Score. The scores are a standardized t-score with mean of 50 and standard deviation of 10.
Peak oxygen utilization (VO2) normalized to weight | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  Peak VO2 will be collected using symptom-limited cardiopulmonary exercise testing (CPET). The average sedentary male will achieve a peak VO2 of approximately 35 to 40 mL/kg/min. The average sedentary female will score a VO2 max of between 27 and 30 mL/kg/min.
Serum Nitrate | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  5 ml of blood will be collected from participants and spun down using a centrifuge to separate the plasma from the rest of the blood. Serological sampling is completed at baseline and at final visit. Serum nitrite (µmol/L) and nitrate levels (µmol/L) will be measured at baseline and after the study intervention to evaluate the successful metabolism of nitrate (in beetroot juice) to nitrite.
VO2 at anaerobic threshold (AT) normalized to weight | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  VO2 (ml/kg/min) at AT will be assessed using symptom-limited CPET. The VO2 at AT for the general population occurs at approximately 50-60% of the peak VO2.
Serum Nitrite | Baseline (pre-intervention) to Follow-up (post-intervention); approx. 2 weeks
  5 ml of blood will be collected from participants and spun down using a centrifuge to separate the plasma from the rest of the blood. Serological sampling is completed at baseline and at final visit. Serum nitrite (µmol/L) and nitrate levels (µmol/L) will be measured at baseline and after the study intervention to evaluate the successful metabolism of nitrate (in beetroot juice) to nitrite.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Forman, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leuenberger AE. [Clinical experience with the O'Malley LOG2 photocoagulator (author's transl)]. Klin Monbl Augenheilkd. 1977 Jan;170(1):143-6. German. PMID 850349
- [Background] Gullis RJ, Rowe CE. Pharmacological studies on the stimulation of the phospholipase A2-acylation system of synaptic membranes of brain, by neurotransmitters and other agonists. J Neurochem. 1976 Jun;26(6):1217-30. doi: 10.1111/j.1471-4159.1976.tb07010.x. No abstract available. PMID 778343 (Retraction: PMID 400955 J Neurochem. 1977 Jun;28(6):1159)
- [Background] Appelboom T, Famaey JP. [Allopurinol and gouty hyperuricemia : apropos of 30 cases treated by a single daily dose]. Brux Med. 1977 Mar;57(3):133-7. No abstract available. French. PMID 861817
- [Background] Westman WE. Problems in implementing U.S. water quality goals. Am Sci. 1977 Mar-Apr;65(2):197-203. No abstract available. PMID 403838
- [Background] Ansehn S, Winblad B. Surface morphology of Candida albicans after treatment with antimycotic drugs. Mykosen Suppl. 1978;1:322-7. No abstract available. PMID 400881
- [Background] Baggiolini M. [The release of proteinases from neutrophil leukocytes and macrophages]. Bull Schweiz Akad Med Wiss. 1979 Sep;35(4-6):283-99. German. PMID 394786
- [Background] Devine CJ Jr, Franz JP, Horton CE. Evaluation and treatment of patients with failed hypospadias repair. Trans Am Assoc Genitourin Surg. 1977;69:4-7. PMID 369094
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Pesta D, Gnaiger E. High-resolution respirometry: OXPHOS protocols for human cells and permeabilized fibers from small biopsies of human muscle. Methods Mol Biol. 2012;810:25-58. doi: 10.1007/978-1-61779-382-0_3. PMID 22057559
- [Background] Vogiatzis I, Zakynthinos S. The physiological basis of rehabilitation in chronic heart and lung disease. J Appl Physiol (1985). 2013 Jul 1;115(1):16-21. doi: 10.1152/japplphysiol.00195.2013. Epub 2013 Apr 25. PMID 23620491
- [Background] Czyzewski K, Pudelski J, Dzielicki J, Guzy R. [Respiratory disorders as a consequence of thoracic injuries]. Pol Przegl Chir. 1979 Jan;51(1):1-6. No abstract available. Polish. PMID 461237
- [Background] Ferguson SK, Woessner MN, Holmes MJ, Belbis MD, Carlstrom M, Weitzberg E, Allen JD, Hirai DM. Effects of inorganic nitrate supplementation on cardiovascular function and exercise tolerance in heart failure. J Appl Physiol (1985). 2021 Apr 1;130(4):914-922. doi: 10.1152/japplphysiol.00780.2020. Epub 2021 Jan 21. PMID 33475460
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Effects of dietary nitrate on oxygen cost during exercise. Acta Physiol (Oxf). 2007 Sep;191(1):59-66. doi: 10.1111/j.1748-1716.2007.01713.x. Epub 2007 Jul 17. PMID 17635415
- [Background] Eggebeen J, Kim-Shapiro DB, Haykowsky M, Morgan TM, Basu S, Brubaker P, Rejeski J, Kitzman DW. One Week of Daily Dosing With Beetroot Juice Improves Submaximal Endurance and Blood Pressure in Older Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):428-37. doi: 10.1016/j.jchf.2015.12.013. Epub 2016 Feb 10. PMID 26874390
- [Background] Hirai DM, Zelt JT, Jones JH, Castanhas LG, Bentley RF, Earle W, Staples P, Tschakovsky ME, McCans J, O'Donnell DE, Neder JA. Dietary nitrate supplementation and exercise tolerance in patients with heart failure with reduced ejection fraction. Am J Physiol Regul Integr Comp Physiol. 2017 Jan 1;312(1):R13-R22. doi: 10.1152/ajpregu.00263.2016. Epub 2016 Oct 26. PMID 27784687
- [Background] Woessner MN, Neil C, Saner NJ, Goodman CA, McIlvenna LC, Ortiz de Zevallos J, Garnham A, Levinger I, Allen JD. Effect of inorganic nitrate on exercise capacity, mitochondria respiration, and vascular function in heart failure with reduced ejection fraction. J Appl Physiol (1985). 2020 May 1;128(5):1355-1364. doi: 10.1152/japplphysiol.00850.2019. Epub 2020 Apr 2. PMID 32240013
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745
- [Background] Forman DE, Arena R, Boxer R, Dolansky MA, Eng JJ, Fleg JL, Haykowsky M, Jahangir A, Kaminsky LA, Kitzman DW, Lewis EF, Myers J, Reeves GR, Shen WK; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Prioritizing Functional Capacity as a Principal End Point for Therapies Oriented to Older Adults With Cardiovascular Disease: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2017 Apr 18;135(16):e894-e918. doi: 10.1161/CIR.0000000000000483. Epub 2017 Mar 23. PMID 28336790
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013

DOCUMENTS (1):
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT05618574/ICF_000.pdf